CLINICAL TRIAL: NCT04599595
Title: Characteristics of INTESTINAL DYSFUNCTION in Patients With MULTIPLE SCLEROSIS. Effectiveness of the TRANSANAL IRRIGATION PROCEDURE With the PERISTEEN DEVICE in the Treatment of Constipation and Disease-related Anal Incontinence
Brief Title: Characteristics of INTESTINAL DYSFUNCTION in Patients With MULTIPLE SCLEROSIS
Status: Completed | Type: Observational
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Simona Ascanelli, Principal Investigator, University Hospital of Ferrara
Other Study IDs: 170485
Record Dates: First submitted 2020-05-23; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Multiple Sclerosis; Intestinal Dysfunction; Anal Incontinence; Microbiota
Keywords: transanal irrigation
MeSH Terms: conditions — Multiple Sclerosis; Encopresis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The faecal sample will be stored at -20 C° and then it will be sent to the Laboratory of the Department of Pharmacy and Biotechnology of the University of Bologna, Italy, for the analysis of the intestinal microbiome composition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Multiple Scerosis (MS) Group: This group will be composed by 150 MS patients who, consecutively, from the start of the study, will refer to the MS clinic of the Neurology Unit of the Ferrara University Hospital, Italy. The first 50 patients with a PACQoL score ≥ 32 will be asked to be willing to enter the next phase of the study that continues at the Coloproctological Outpatient Clinic of Ferrara University Hospital, Italy with an appointment provided by the neurologist with a pre-established schedule (with written consent).
  Interventions: Device: Peristeen (Coloplast)

INTERVENTIONS:
Device: Peristeen (Coloplast) — Patients with severe intestinal dysfunction impairment (PAC QoL score ≥ 32) will be offered the adoption of the TAI (Transanal Irrigation) with Peristeen Device as a way to manage their own evacuation, replacing any other measure used until that moment (suppositoires, clisms exceptionally cc) with the exception of the possible intake of macrogols and/or prebiotics and/or probiotics which instead patients can continue. This treatment will be proposed to all patients with severe impairment of intestinal function.
  The TAI training with Peristeen will be carried out at the surgical clinic of the Surgical Department of the Ferrara University Hospital, Italy, by the health personnel involved in the study, usually in a single session, but more sessions may be necessary, with the continuation of the TAI for 4 weeks or with patient's exclusion from the study if the guarantees of appropriate use of the device will not be reached.

SUMMARY:
MS (Multiple Sclerosis) is the most common neurological disease involving disabilities in young adults, with bowel symptoms, in particular constipation and fecal incontinence. The main objectives of the study are to assess the prevalence, characteristics, severity and impact on the Quality of Life of intestinal disorders in this population, to correlate the severity and characteristics of constipation and fecal incontinence with Intestinal Transit Time and the time dedicated to the evacuation, and how these items change in relation to the use of transanal irrigation (TAI). Another objective is to identify the composition of the intestinal microbiota in MS patients in relation to the type of bowel characteristics, comparing it with microbiota profile of the healthy population of the same region of origin, Emilia-Romagna, Italy.

DETAILED DESCRIPTION:
MS (Multiple Sclerosis) is the most common neurological disease involving disabilities in young adults, with Central Nervous System involvement in both the brain and spinal cord. In a recent review, its incidence in the United Kingdom is estimated at 7 new cases per 100,00 inhabitants per year, with a prevalence of about 100,000 patients. Bowel symptoms, in particular constipation and faecal incontinence, affect more than two thirds of MS patients, and have a significant impact on patients' quality of life (QoL) by significantly limiting their social, occupational and emotional life.

Recently, bowel management based on Transanal Irrigation (TAI) has also been proposed in patients with MS, but TAI efficacy on intestinal transit time and patient's compliance with TAI have not been defined yet.

The primary objective of the study is to assess the prevalence, characteristics, severity and impact on the Quality of Life of intestinal disorders in patients who consecutively refer to the neurological clinic for the diagnosis and treatment of Multiple Sclerosis at Ferrara University Hospital, Italy.

Secondary objectives are to correlate the severity and characteristics of constipation and fecal incontinence with intestinal transit time and the type of faeces evacuated according to the Bristol Stool Form Scale; to evaluate the costs in terms of the precautions (diapers, traverses, drugs, medicated clysms, etc.) and the time dedicated to the evacuation, and how these items change in relation to the use of TAI; and finally, to study the composition of the intestinal microbiota in MS patients in relation to the type of bowel characteristics, comparing it with the profile of the healthy population of the same region of origin, Emilia-Romagna, Italy.

The study proposed is a monocentric prospective observational study. The study population will be composed of patients who will consecutively refer to the Neurological Clinics of the University Hospital of Ferrara, Italy for a number of about 150 patients.

The study will consist of two phases.The first phase will be the selection of eligible patients by administering two self-filling questionnaires: PacQol (Patient Assessment of Constipation Quality of Life) and NBD (Neurogenic Bowel Dysfunction Score).

Patients with PacQol score ≥ 32 will be sent to the surgical clinic for the second phase. During the latter phase, patients will undergo a number of visits varying from 1 to 4 depending on the patient's willingness to continue the study. After the illustration of the purpose and protocol of the study to the patient, classification of constipation and/or faecal incontinence in accordance with the Rome III Diagnostic Criteria will be assessed, with consideration of other possible etiopathogenetic factors other than MS. Further questionnaires will be filled in to evaluate the disease status (Constipation scoring system by Agachan-Wexner, Obstructed defecation score by Altomare, Fecal Incontinente grading scale by Jorge-Wexner); if the patient will consent to the continuation of the study, he will be given 7-days food diaries, evacuation diaries, radiopaque markers, stool collection container and appointment date for plain abdominal X-ray which may coincide with the appointment for examination number 2 (visit 2 or 3).

In particular, radiopaque markers Intestinal Transit Study will be performed according to the Bouchoucha procedure revised by Abrahamsson, which involves ingestion of 10 markers for 6 days at the same time and execution of a plain abdominal X-ray on the 7th day. During this week the patient will complete an evacuation diary recording the time and number of evacuations, the method of eventual bowel care, the consistency of faeces according to the Bristol Scale, any episode of fecal incontinence, the type of hygiene measures in general, the number of enemas, diapers, and any other garrison used in relation to the evacuation.

Patients will be asked to collect a faecal sample in a container during the last week before the following inspection at Visit 2.

During the second visit, the outcome of the plain abdominal X-ray will be discussed, the completed diaries will be collected, and the faecal sample will be stored at -20 C° and subsequentely sent to the Laboratory of the Department of Pharmacy and Biotechnology of the University of Bologna, Italy for the analysis of the intestinal microbiome composition.

Patients with severe NBD impairment will be offered the adoption of TAI as a way to manage their own evacuation, replacing any other measure used until that moment (suppositoires, enemas) with the exception of the possible intake of macrogols and/or prebiotics and/or probiotics which instead can be continued. This treatment will be proposed to all patients with severe impairment of intestinal function.

The TAI training with Peristeen will be carried out at the surgical clinic of the Surgical Department of the Ferrara University Hospital, Italy, by the personnel involved in the study, usually in a single session, but more sessions may be necessary.

During the following 4 weeks, patients will continue to use the Peristeen at home according to the instructions provided by the training staff collecting a stool sample each week. During the last of the four weeks of TAI use patients will repeat the compilation of food diaries, evacuation diaries, the radiopaque markers Transit Time, and collection of the stool for microbiota analysis. The appointment for the radiography could coincide also in this case with the following visit (visit 3 or 4).

During the last visit the outcome of Transit Time X-ray will be discussed, completed diaries and stool samples will be collected, and PAC-QoL questionnaire will be submitted to patients who completed the study pathway.

Patients will be asked about overall satisfaction of TAI treatment with Peristeen by means of a numerical assessment from 0 to 10.

Finally, any comment will be noted as well any events that might be related to TAI irrigation with Peristeen will be recorded.

Patients will undergo a neurological examination 3 months after the start of treatment.

The whole duration of the study will be of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age, both sexes
* Diagnosis of MS for no more than 10 years
* Residence in the Italian Region of Emilia Romagna, Italy

Exclusion Criteria:

* EDSS (Expanded Disability Status Scale) < or =7
* Diagnosis of Celiac Disease, Inflammatory Bowel Disease (Ulcerative Colitis or Crohn's Disease)
* Evidence of Diverticular Colon Disease
* Previous or ongoing neoplastic diseases of the digestive system
* Endocrine disorders such as uncompensated hypothyroidism, diabetes mellitus in treatment, hypoparathyroidism, pheochromocytoma
* Other neurological disorders such as M. of Parkinson's, S. of Shy Drager.
* Taking drugs that affect intestinal transit (opiates, antiepileptic drugs, major antidepressants, calcium antagonists, anticholinergics, antidopaminergics)
* Evidence of rectal or occult bleeding in the last 3 months
* Infectious episodes in progress (*)

NOTES:

(*) Rational: it is not considered ethical or functional to carry out such research in patients with infectious organ diseases requiring antibiotic and/or inflammatory therapies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be composed by 150 MS patients who will consecutively refer to the MS Outpatient Neurology Clinic at Ferrara University Hospital, Italy. The PAC-QoL questionnaire will be given to every patient. This questionnaire is a self-filled instrument validated and used in various studies to document the consequences that intestinal disorders and defecation have on everyday life. The first 50 patients with a PACQoL score ≥ 32 will be asked to be willing to enter the next phase of the study that continues at the Coloproctological Outpatient Clinic of Ferrara University Hospital, Italy with an appointment provided by the neurologist with a pre-established schedule (with written consent).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2020-04-10 (Actual)

PRIMARY OUTCOMES:
Incidence and prevalence of intestinal dysfunction in Multiple sclerosis | 2 years
  Incidence and prevalence of intestinal dysfunction in Multiple Sclerosis by calculation of percentage of patients with a PACQoL score ≥ 32 for items B.1 to B.6 and/or a score ≤ 11 for item B.7 of the questionnaire.
Intestinal transit time in SM patients with intestinal dysfunction | 2 years
  Calculation of percentage of patients with a slowed Intestinal Transit Time (≥ 60 hours for females and 55 hours for men)

SECONDARY OUTCOMES:
Analysis of Microbiota in MS patients with intestinal dysfunction, before and after treatment with TAI. | 2 years
  Compare the composition of the intestinal microbiota of MS patients with the known "healthy" profile of the Italian population of North East of Italy and assess any changes after the period of treatment with TAI.

CONTACTS AND LOCATIONS:
Overall Officials: Simona Ascanelli, Principal Investigator — University Hospital of Ferrara
Locations (1):
- Simona Ascanelli, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Koutsouraki E, Costa V, Baloyannis S. Epidemiology of multiple sclerosis in Europe: a review. Int Rev Psychiatry. 2010;22(1):2-13. doi: 10.3109/09540261003589216. PMID 20233110
- [Result] Nordenbo AM, Andersen JR, Andersen JT. Disturbances of ano-rectal function in multiple sclerosis. J Neurol. 1996 Jun;243(6):445-51. doi: 10.1007/BF00900497. PMID 8803816
- [Result] Chia YW, Fowler CJ, Kamm MA, Henry MM, Lemieux MC, Swash M. Prevalence of bowel dysfunction in patients with multiple sclerosis and bladder dysfunction. J Neurol. 1995 Jan;242(2):105-8. doi: 10.1007/BF00887825. PMID 7707085
- [Result] Norton C, Chelvanayagam S. Bowel problems and coping strategies in people with multiple sclerosis. Br J Nurs. 2010 Feb 25-Mar 10;19(4):220, 221-6. doi: 10.12968/bjon.2010.19.4.46783. PMID 20220671
- [Result] Hornby A. The MS sufferer in the community. Nurs Times. 1978 May 11;74(19):suppl 130-1. No abstract available. PMID 652561
- [Result] Nortvedt MW, Riise T, Frugard J, Mohn J, Bakke A, Skar AB, Nyland H, Glad SB, Myhr KM. Prevalence of bladder, bowel and sexual problems among multiple sclerosis patients two to five years after diagnosis. Mult Scler. 2007 Jan;13(1):106-12. doi: 10.1177/1352458506071210. PMID 17294618
- [Result] Wiesel PH, Norton C, Glickman S, Kamm MA. Pathophysiology and management of bowel dysfunction in multiple sclerosis. Eur J Gastroenterol Hepatol. 2001 Apr;13(4):441-8. doi: 10.1097/00042737-200104000-00025. PMID 11338078
- [Result] Preziosi G, Raptis DA, Storrie J, Raeburn A, Fowler CJ, Emmanuel A. Bowel biofeedback treatment in patients with multiple sclerosis and bowel symptoms. Dis Colon Rectum. 2011 Sep;54(9):1114-21. doi: 10.1097/DCR.0b013e318223fd7b. PMID 21825891
- [Result] Wiesel PH, Norton C, Roy AJ, Storrie JB, Bowers J, Kamm MA. Gut focused behavioural treatment (biofeedback) for constipation and faecal incontinence in multiple sclerosis. J Neurol Neurosurg Psychiatry. 2000 Aug;69(2):240-3. doi: 10.1136/jnnp.69.2.240. PMID 10896701
- [Result] Christensen P, Bazzocchi G, Coggrave M, Abel R, Hultling C, Krogh K, Media S, Laurberg S. A randomized, controlled trial of transanal irrigation versus conservative bowel management in spinal cord-injured patients. Gastroenterology. 2006 Sep;131(3):738-47. doi: 10.1053/j.gastro.2006.06.004. PMID 16952543
- [Result] Del Popolo G, Mosiello G, Pilati C, Lamartina M, Battaglino F, Buffa P, Redaelli T, Lamberti G, Menarini M, Di Benedetto P, De Gennaro M. Treatment of neurogenic bowel dysfunction using transanal irrigation: a multicenter Italian study. Spinal Cord. 2008 Jul;46(7):517-22. doi: 10.1038/sj.sc.3102167. Epub 2008 Mar 4. PMID 18317488
- [Result] Bazzocchi G., Poletti E., Avogadri A. L'irrigazione retrograda transanale per il bowel management del paziente con lesione midollare mediante dispositivi a pressione costante, razionale e procedura per l'utilizzo del Peristeen. Pelviperineology 2012; 31: 85-92.
- [Result] Christensen P, Krogh K. Transanal irrigation for disordered defecation: a systematic review. Scand J Gastroenterol. 2010 May;45(5):517-27. doi: 10.3109/00365520903583855. PMID 20199336
- [Result] Emmanuel AV, Krogh K, Bazzocchi G, Leroi AM, Bremers A, Leder D, van Kuppevelt D, Mosiello G, Vogel M, Perrouin-Verbe B, Coggrave M, Christensen P; Members of working group on Trans Anal Irrigation from UK, Denmark, Italy, Germany, France and Netherlands. Consensus review of best practice of transanal irrigation in adults. Spinal Cord. 2013 Oct;51(10):732-8. doi: 10.1038/sc.2013.86. Epub 2013 Aug 20. PMID 23958927
- [Result] Marquis P, De La Loge C, Dubois D, McDermott A, Chassany O. Development and validation of the Patient Assessment of Constipation Quality of Life questionnaire. Scand J Gastroenterol. 2005 May;40(5):540-51. doi: 10.1080/00365520510012208. PMID 16036506
- [Result] Yiannakou Y, Piessevaux H, Bouchoucha M, Schiefke I, Filip R, Gabalec L, Dina I, Stephenson D, Kerstens R, Etherson K, Levine A. A randomized, double-blind, placebo-controlled, phase 3 trial to evaluate the efficacy, safety, and tolerability of prucalopride in men with chronic constipation. Am J Gastroenterol. 2015 May;110(5):741-8. doi: 10.1038/ajg.2015.115. Epub 2015 Apr 14. PMID 25869393
- [Result] Cadeddu F, Salis F, De Luca E, Ciangola I, Milito G. Efficacy of biofeedback plus transanal stimulation in the management of pelvic floor dyssynergia: a randomized trial. Tech Coloproctol. 2015 Jun;19(6):333-8. doi: 10.1007/s10151-015-1292-7. Epub 2015 Mar 6. PMID 25744688
- [Result] Neri L, Basilisco G, Corazziari E, Stanghellini V, Bassotti G, Bellini M, Perelli I, Cuomo R; LIRS Study Group. Constipation severity is associated with productivity losses and healthcare utilization in patients with chronic constipation. United European Gastroenterol J. 2014 Apr;2(2):138-47. doi: 10.1177/2050640614528175. PMID 24953097
- [Result] Bharucha AE, Wald A, Enck P, Rao S. Functional anorectal disorders. Gastroenterology. 2006 Apr;130(5):1510-8. doi: 10.1053/j.gastro.2005.11.064. PMID 16678564
- [Result] Agachan F, Chen T, Pfeifer J, Reissman P, Wexner SD. A constipation scoring system to simplify evaluation and management of constipated patients. Dis Colon Rectum. 1996 Jun;39(6):681-5. doi: 10.1007/BF02056950. PMID 8646957
- [Result] Altomare DF, Spazzafumo L, Rinaldi M, Dodi G, Ghiselli R, Piloni V. Set-up and statistical validation of a new scoring system for obstructed defaecation syndrome. Colorectal Dis. 2008 Jan;10(1):84-8. doi: 10.1111/j.1463-1318.2007.01262.x. Epub 2007 Apr 18. PMID 17441968
- [Result] Jorge JM, Wexner SD. Etiology and management of fecal incontinence. Dis Colon Rectum. 1993 Jan;36(1):77-97. doi: 10.1007/BF02050307. PMID 8416784
- [Result] Krogh K, Christensen P, Sabroe S, Laurberg S. Neurogenic bowel dysfunction score. Spinal Cord. 2006 Oct;44(10):625-31. doi: 10.1038/sj.sc.3101887. Epub 2005 Dec 13. PMID 16344850
- [Result] Bouchoucha M, Devroede G, Arhan P, Strom B, Weber J, Cugnenc PH, Denis P, Barbier JP. What is the meaning of colorectal transit time measurement? Dis Colon Rectum. 1992 Aug;35(8):773-82. doi: 10.1007/BF02050328. PMID 1644002
- [Result] Abrahamsson H, Antov S. Accuracy in assessment of colonic transit time with particles: how many markers should be used? Neurogastroenterol Motil. 2010 Nov;22(11):1164-9. doi: 10.1111/j.1365-2982.2010.01543.x. PMID 20584262

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-06-29): https://cdn.clinicaltrials.gov/large-docs/95/NCT04599595/Prot_SAP_000.pdf
  • Informed Consent Form (2017-06-29): https://cdn.clinicaltrials.gov/large-docs/95/NCT04599595/ICF_001.pdf